CLINICAL TRIAL: NCT05951179
Title: A Phase 2, Open-Label Study to Evaluate the Safety and Efficacy of Intravesical Instillation of TARA-002 in Adults With High-Grade Non-Muscle Invasive Bladder Cancer
Brief Title: Safety and Efficacy Study of Intravesical Instillation of TARA-002 in Adults With High-grade Non-muscle Invasive Bladder Cancer
Acronym: ADVANCED-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Protara Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TARA-002-101-Ph2
Record Dates: First submitted 2023-06-29; First posted 2023-07-18 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Non-muscle Invasive Bladder Cancer
Keywords: Non-muscle invasive bladder Cancer; bladder cancer; high grade Ta; high grade NMIBC; carcinoma in situ
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms; Carcinoma in Situ

STUDY DESIGN:
Intervention Model Description: All participants will receive 6 weekly instillations of TARA-002 at the established RP2D (First Treatment Period). Participants who are eligible for reinduction after the First Treatment Period will receive 6 additional weekly doses of TARA-002 instillation as part of the Second Treatment Period. Participants confirmed to have a complete response after the First Treatment Period will receive 3 additional weekly doses of TARA-002 instillation as maintenance during the Second Treatment Period. All eligible participants will receive 3 weekly doses of TARA-002 instillation as part of the Third Treatment Period (maintenance) at Months 6, 9, 12, 15,18, and 24. Following the Third Treatment Period, all participants will continue to the Follow up Period from Month 27 until Month 60.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TARA-002 (Experimental): TARA-002 is a lyophilized biological preparation for instillation containing cells of Streptococcus pyogenes (Group A, type 3) Su strain.
  Interventions: Biological: TARA-002

INTERVENTIONS:
Biological: TARA-002 — All participants will receive 6 weekly instillations of TARA-002 at the established RP2D (First Treatment Period). Participants who are eligible for reinduction after the First Treatment Period will receive 6 additional weekly doses of TARA-002 instillation as part of the Second Treatment Period. Participants confirmed to have a complete response after the First Treatment Period will receive 3 additional weekly doses of TARA-002 instillation as maintenance during the Second Treatment Period. All eligible participants will receive 3 weekly doses of TARA-002 instillation as part of the Third Treatment Period (maintenance) at Months 6, 9, 12, 15, and 18. Following the Third Treatment Period, all participants will continue to the Follow up Period from Month 21 until Month 60.

SUMMARY:
TARA-002-101-Ph2 is an open-label study to investigate the safety and efficacy of intravesical instillation of TARA-002 in adults 18 years of age or older with high-grade CIS NMIBC (± Ta/T1).

The purpose of this Phase 2 study (TARA-002-101-Ph2) is to further assess the safety and efficacy of TARA-002 at the RP2D which has been established in the Phase 1a dose finding study (TARA-002-101-Ph1a).

This Phase 2 study includes participants with CIS NMIBC (± Ta/T1) with active disease, defined as disease present at last tumor evaluation (within 3 months) prior to signing the ICF.

Participants will be enrolled into one of 2 cohorts:

Cohort A:

* Participants with CIS (± Ta/T1) who are BCG naive, or
* Participants with CIS (± Ta/T1) who are BCG exposed and have not received intravesical BCG for at least 24 months prior to the most recent CIS diagnosis

Cohort B:

* Participants who are BCG unresponsive

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants 18 years of age or older at the time of signing informed consent
* Participants who have voluntarily given written informed consent after the nature of the study has been explained according to applicable requirements prior to study entry
* Central histologic confirmation of high-grade non-muscle invasive CIS (± Ta/T1) with active disease
* Participants who are BCG naive, or participants who are BCG exposed and have not received intravesical BCG for at least 24 months prior to the most recent CIS diagnosis (Cohort A). Participants with CIS (± Ta/T1) who are BCG unresponsive.

Exclusion Criteria:

* Penicillin allergy (participants with a questionable history of allergy to penicillin will undergo penicillin blood allergy testing via central laboratory
* Central confirmed variant histology
* Concomitant prostatic or upper tract urothelial involvement per Investigator's assessment
* Nodal and metastatic disease are excluded if they existed at any time (whether present or in the past)
* Any history of ≥ T2 bladder cancer that existed at any point in time in the participant's history

For more information on eligibility criteria, please contact the Sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2030-05 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Cohort A and B: Incidence of high-grade Complete Response at any time according to central pathology after treatment with TARA-002 | Month 3 to Month 60
Cohort A: Incidence of high-grade Complete Response at any time by subgroup (BCG naive and BCG exposed > 24 months) according to central pathology after treatment with TARA-002 | Month 3 to Month 60

SECONDARY OUTCOMES:
Cohort A and B: Duration of high-grade Complete Response rate at Months 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 36, 42, 48, 54, and 60 after treatment with TARA-002 | Month 3 to Month 60
Cohort A and B: High-grade Complete Response rate at Months 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 36, 42, 48, 54, and 60 after treatment with TARA-002 | Month 3 to Month 60
Cohort A and B: Duration of Complete Response (all recurrent bladder cancer, including low grade Ta) after treatment with TARA-002 | Month 3 to Month 60
Cohort A and B: Complete Response rate (all recurrent bladder cancer, including low grade Ta) at Months 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 36, 42, 48, 54, and 60 after treatment with TARA-002 | Month 3 to Month 60
Cohort A and B: Progression free survival after treatment with TARA-002 | 60 months
Cohort A and B: Disease-specific progression free survival after treatment with TARA-002 | 60 months
Cohort A and B: Overall survival after treatment with TARA-002 | 60 months
Cohort A and B: Disease specific survival after treatment with TARA-002 | 60 months
Cohort A and B: Time to cystectomy after treatment with TARA-002 | 60 months
Cohort A and B: Time to recurrence delayed cystectomy after treatment with TARA-002 | 60 months
Cohort A and B: Time to progression after treatment with TARA-002 | 60 months
Cohort A and B: Time to disease worsening after treatment with TARA-002 | 60 months
Cohort A and B: Incidence and severity of AEs, TEAEs, SAEs and TESAEs after treatment with TARA-002 | Day 1 to Month 60
  AE = adverse event; TEAE = treatment emergent adverse event; SAE = serious adverse event; TESAE = treatment emergent serious adverse event
Cohort A and B: Change from baseline in urine pharmacodynamic biomarker levels (including IL-6, IL-8, IFN-γ, and TNF-α) after treatment with TARA-002 | Day 1 to Day 72
Cohort A and B: Quality of Life based on the EORTC questionnaire QLQ-NMIBC24 | Day 1 to Month 24
  EORTC = European Organization for Research and Treatment of Cancer; QLQ-NMIBC24 = Questionnaire for Patients with NMIBC
Cohort A and B: Quality of Life based on the EORTC questionnaire QLQ-C30 | Day 1 to Month 24
  EORTC = European Organization for Research and Treatment of Cancer; QLQ-C30 = Questionnaire for Patients with Cancer

CONTACTS AND LOCATIONS:
Overall Officials: Chief Scientific Operations Officer, Study Director — Protara Therapeutics
Locations (61):
- United States (38):
  - Urology Centers of Alabama, Homewood, Alabama
  - Mayo Clinic, Phoenix, Arizona
  - East Valley Urology Center of Arizona, Queen Creek, Arizona
  - Arkansas Urology, Little Rock, Arkansas
  - Michael Oefelein Clinical Trials, Bakersfield, California
  - Urology Group of Southern California, Los Angeles, California
  - University of California Irvine Medical Center, Orange, California
  - Genesis Research, San Diego, California
  - Genesis Research LLC, Torrance, California
  - Colorado University - Anshutz, Aurora, Colorado
  - AdventHealth Medical Group Urology of Denver, Denver, Colorado
  - Advanced Urology, Lakewood, Colorado
  - Urology Associates of Denver, Lone Tree, Colorado
  - University of Florida Health Jacksonville, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Comprehensive Urologic Care, Lake Barrington, Illinois
  - Southern Urology, Lafayette, Louisiana
  - Ochsner Health LSU - Regional Urology, Shreveport, Louisiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Specialty Clinic Research of St. Louis, St Louis, Missouri
  - AccuMed Research Associates, Garden City, New York
  - University of Rochester, Department of Urology, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of Toledo, Toledo, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Conrad Person Clinic, Memphis, Tennessee
  - Urology Associates PC, Nashville, Tennessee
  - Amarillo Urology Research, Amarillo, Texas
  - Urology Partners of North Texas, Arlington, Texas
  - Urology Austin, LLC, Austin, Texas
  - Houston Metro Urology, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - UT Health San Antonio, San Antonio, Texas
  - Virginia Urology, Richmond, Virginia
- Argentina (5):
  - Centro Argentino de Urologia, CABA
  - Hospital Sirio Libanes, CABA
  - Centro Urologico Profesor Bengio SA, Córdoba
  - CEMAIC, Córdoba
  - Clinica Privada Independencia, Munro
- Brazil (10):
  - Fuji City General Hospital, Nova Lima, Minas Gerais
  - Kyushu University Hospital, Nova Lima, Minas Gerais
  - Office of Lucas Nougeria MA, Nova Lima, Minas Gerais
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Nucleo de Pesquisa Clinica do Rio Grande so Sul, Porto Alegre, Rio Grande do Sul
  - Centro de Urologia Avancada, Porto Alegre, Rio Grande do Sul
  - Komaki City Hospital, Porto Alegre, Rio Grande do Sul
  - Hospital de Clinicas da UNICAMP, Campinas, São Paulo
  - Instituto Dor de Pesquisa e Ensino, Jardim Paulista, São Paulo
  - Faculdade de Medicina ABC-CEPHO, Santo André, São Paulo
- Canada (4):
  - Exdeo Clinical Research Inc, Abbotsford, British Columbia
  - Jonathan Giddes Medicine Professional Corporation, Brampton, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - UHN Princess Margaret Cancer Centre Princess Margaret Hospital, Toronto, Ontario
- Japan (3):
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Japanese Red Cross Osaka Hospital, Osaka, Osaka
  - Tokyo University Medical Center Sakura Hospital, Fuji-shi, Shizuoka
- Arensia Kapitanivka - PPDS, Kapitanivka, Ukraine

IPD SHARING:
Plan to Share IPD: No